CLINICAL TRIAL: NCT05994703
Title: Assisting Smokers to Switch to an e-Cigarette by Accelerating Learning of Adaptive Habits Using D-cycloserine
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Rose Research Center, LLC (Industry)
Collaborators: Foundation for a Smoke Free World INC (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CYCLE
Record Dates: First submitted 2023-07-24; First posted 2023-08-16 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Smoking Cessation; Harm Reduction
MeSH Terms: conditions — Smoking Cessation; Harm Reduction | interventions — Cycloserine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- DCS with Juul e-cigarette (Experimental): d-cycloserine (DCS) 100 mg taken orally, once a day for six weeks. There will be a 50 mg dose taken the afternoon/evening prior to the first switch date (after enrollment) to ensure serum levels of the medication are available for the first switch to e-cigarette attempt.
  Participants will be instructed to use the Juul as often as they like during the 12 week period, and to switch completely to the Juul within 1 week. If, however, they do smoke any combustible cigarettes (CC), they will also be instructed to use the Juul immediately before each CC to relieve their craving as much as possible before smoking their usual brand. The Juul will also be the first product that they are instructed to use each morning. Smokers will be told to try to completely substitute Juul for CCs by the end of the first week of use.
  Interventions: Drug: d-cycloserine; Other: Juul e-cigarette

INTERVENTIONS:
Drug: d-cycloserine — d-cycloserine (DCS) 100 mg taken orally, once a day for six weeks.
Other: Juul e-cigarette — Juul use as often as the participant likes for 12 weeks.

SUMMARY:
This study will evaluate the effects of a reward devaluation strategy, which has been researched in the past, combined/augmented with the medication d-cycloserine in assisting smokers to switch from combustible cigarette (CC) to Juul.

ELIGIBILITY:
Inclusion Criteria:

1. Has signed the informed consent form (ICF) and is able to understand the information provided in the ICF.
2. Is 22 to 65 years of age (inclusive) at screening.
3. Smokes ≥ 10 commercially available CCs per day (no brand restrictions), for the last 12 months.
4. Expired air CO reading of at least 10 ppm as assessed at the screening session.
5. Interested in switching to an electronic cigarette.
6. Willing and able to comply with the requirements of the study.
7. Owns a smart phone with text message and data capabilities compatible with necessary surveys.

Exclusion Criteria:

1. Is unhealthy or cannot participate in the study for any reason (e.g., medical, psychiatric, and/or social reason) as judged by the Investigator or designated medical staff based on all available assessments from the screening period (e.g., safety laboratory, vital signs, physical examination, ECG, concomitant medications and medical history).
2. Patient Health Questionnaire (PHQ-9) score greater than 9, or a score greater than 0 on item #9 ("Thoughts that you would be better off dead, or of hurting yourself in some way") at screening.
3. Planned use of an FDA-approved smoking cessation product during the study.
4. High Blood Pressure (systolic >150 mm Hg, diastolic >95 mm Hg) at screening.
5. Body mass index (BMI) less than 15.0 kg/m2 or greater than 40.0 kg/m2.
6. Coronary heart disease, structural cardiac disease (including, but not limited to valvular heart disease or cardiac murmurs), cardiac dysrhythmias, syncope, cardiac chest pain, or history of heart attack or heart failure.
7. Has received psychotherapy or behavioral treatments within 30 days of screening, or during the study.
8. Taking antidepressants or psychoactive medications (e.g., antipsychotics, antidepressants, benzodiazepines, hypnotics).
9. Use of any of these products in the past 30 days:

   1. Illegal drugs (or if the urine drug screen is positive for cocaine, tetrahydrocannabinol (THC), amphetamines, methamphetamines, or opiates);
   2. Experimental (investigational) drugs that are unknown to participant;
   3. Chronic opiate use;
   4. Medications to treat tuberculosis (e.g., isoniazid, ethionamide).
10. Use of smokeless tobacco (chewing tobacco, snuff), cigars (except for "Black & Mild" cigars or Cigarillos), pipes, hookah, e-cigarettes, nicotine replacement therapy or other smoking cessation treatments within 14 days of screening.
11. Pregnant or nursing (by self-report) or positive pregnancy test.

Ages: 22 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2023-10-20 (Actual); Primary Completion 2025-10-13 (Actual); Study Completion 2026-01-12 (Actual)

PRIMARY OUTCOMES:
Smoking Abstinence based on Self-Report | During weeks 3-6 and 9-12 post-switching date.
  Complete switching from combustible cigarette use at each time point will be defined by a self-report of no cigarette smoking (not even a puff) since the prior session.
Smoking Abstinence based on Expired Air Carbon Monoxide (CO) | End of Week 6, End of Week 12
  Complete switching from combustible cigarette use at each time point will be confirmed by an expired air CO reading of less than 5 ppm.

SECONDARY OUTCOMES:
Reduction in Cigarettes Per Day | Week 6, Week 12, Six-Month Follow-Up
  Reduction in the number of reports cigarettes smoked per day over the previous seven days (at each time point) compared to baseline.
Reduction in Expired Air Carbon Monoxide (CO) | End of Week 6, End of Week 12
  Reduction in Expired Air Carbon Monoxide (CO) compared to baseline.
Change in rewarding effects for cigarettes and e-cigarettes at 6 weeks post switch | End of Week 6
  o assess subjective satisfaction and other perceived rewarding or aversive effects accompanying e-cigarette use and combustible cigarette use using the modified (e-Cigarette) Cigarette Evaluation Questionnaire. This questionnaire contains five subscale scores: smoking satisfaction (satisfying, tastes good, enjoy smoking), psychological rewards (calms down, more awake, less irritable, helps concentrate, reduces hunger), aversion (dizziness, nauseated), enjoyment of respiratory tract sensations (single-item assessment), craving reduction (single-item assessment). Participants will be asked to assess the 12 items of the questionnaire on a 7-point scale, ranging from "1-not at all" to "7-extremely".

OTHER OUTCOMES:
Tolerability of daily use of D-cycloserine in conjunction with Juul | Week 2, Week 6, Week 8, Week 12
  The frequency and severity of adverse events will be tabulated as well as the likelihood of their causal relationship to treatment.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Rose Research Center, Charlotte, North Carolina
  - Rose Research Center, Raleigh, North Carolina

IPD SHARING:
Plan to Share IPD: No